CLINICAL TRIAL: NCT03649087
Title: Testing of Vitrification Protocols for Ovarian Tissue Harvesting in Female to Male Transsexuals
Brief Title: Vitrification for Ovarian Tissue Harvesting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maximilian Franz, M.D. (Other)
Responsible Party: Sponsor-Investigator, Maximilian Franz, M.D., MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2204
Record Dates: First submitted 2017-10-29; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Ovary; Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Vitrification

STUDY DESIGN:
Intervention Model Description: Vitrification of ovarian tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vitrification — Vitrification of ovarian tissue

SUMMARY:
Increasing interest has emerged concerning ovarian tissue cryopreservation and subsequent transplantation as a potential way of preserving fertility in cancer patients as well as for women who just wish to delay childbearing. As the majority of existing protocols use the slow freezing method, this study aims to test vitrification techniques of ovarian cortex.

ELIGIBILITY:
Inclusion Criteria:

* female-to-male transsexuals
* gender completing operation
* signed informed consent form
* willingness to donate ovarian tissue for research purposes
* age >=18 years

Exclusion Criteria:

* malignant disease
* age under 18 years
* refusal to donate ovarian tissue

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female-to-male transsexuals
Enrollment: 10 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
survival of ovarian tissue | 2 days until 2 years after freezing
  histologic and enzymatic evaluation of ovarian tissue with respect to survival and functionality of ovarian follicles

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Obstetrics and Gynaecology of the Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marschalek J, Egarter C, Nouri K, Dekan S, Ott J, Frank M, Pietrowski D. The effect of different vitrification protocols on cell survival in human ovarian tissue: a pilot study. J Ovarian Res. 2021 Dec 6;14(1):170. doi: 10.1186/s13048-021-00924-8. PMID 34872604
- [Derived] Marschalek J, Pietrowski D, Dekan S, Marschalek ML, Brandstetter M, Ott J. Markers of vitality in ovaries of transmen after long-term androgen treatment: a prospective cohort study. Mol Med. 2020 Sep 5;26(1):83. doi: 10.1186/s10020-020-00214-x. PMID 32891132